CLINICAL TRIAL: NCT05205642
Title: The Evaluation of Exercise Fatigue Parameters and Endothelial Function in Pediatric Patients With a History of COVID-19 Infection or Multisystem Inflammatory Syndrome (MIS-C)
Brief Title: Exercise Fatigue Parameters and Endothelial Function in Pediatric Patients With a History of COVID-19 Infection or MIS-C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0768-20-RMB
Record Dates: First submitted 2022-01-23; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; MIS-C Associated With COVID-19
Keywords: Cardiopulmonary Exercise Testing; EndoPAT; COVID-19
MeSH Terms: conditions — COVID-19; pediatric multisystem inflammatory disease, COVID-19 related | interventions — Exercise Test

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients recovering from COVID-19 (Experimental): Pediatric and adult patients recovering from COVID-19 with or without complaints.
  Interventions: Device: Cardiopulmonary exercise test (CPET); Device: Peripheral Arterial Tonography (PAT) using the EndoPAT™ device; Diagnostic Test: Endothelin

INTERVENTIONS:
Device: Cardiopulmonary exercise test (CPET) — Cardiopulmonary exercise testing (CPET) using a Quark CPET metabolic cart (Rome, Italy) according to American Thoracic Society (ATS) guidelines. A symptom-limited test on a treadmill will be performed, using incremental ramp Bruce protocol up to exhaustion. Patients who will not be able to perform the test on a treadmill will be tested on a cycle ergometer beginning with a no-resistance warm-up lasting 2-3 minutes, followed by incrementing resistance (8-30 Watts/minute) adapted to the patient's functional capacities according to the examiner's free judgment, up to exhaustion.
Device: Peripheral Arterial Tonography (PAT) using the EndoPAT™ device — A volume sensor measuring reactive hyperemia is placed on the second fingertip of both hands. First the device evaluates the baseline volume of the pulse. Then, we will apply pressure that is 50 mmHg higher than the baseline systolic pressure of the examinee on the evaluated hand for five minutes, using a sphygmomanometer cuff. After the pressure is released on the evaluated hand, the new pulse volume is tested. To neutralize the effects of the autonomous systemic response, the program divides the difference of the pulse volume in the examined hand by the difference in the untested hand and we get the Reactive Hyperemic Index (RHI) which represents the endothelial function in the tested hand. During the examination, the calculated arterial tonometry graph is generated, and out of it the RHI will be automatically calculated, using the EndoPAT2000™ program.
Diagnostic Test: Endothelin — For Endothelin levels we will use the Endothelin ELISA kit from R&D company, and for measurement 1 cc of serum will be needed.

SUMMARY:
Acute coronavirus disease 2019 (COVID-19) infection can include cardiac and pulmonary manifestations as well as post-infectious complications such as multisystem inflammatory syndrome (MIS-C), also known as pediatric inflammatory multisystem syndrome (PIMS / PIMS-TS). The precise etiology for COVID-19 symptoms and MIS-C is still obscure but there is evidence that endothelial damage may play a role. At recovery, symptoms such as dyspnea, fatigue, weakness, myalgia, chest pain and palpitations are prevalent. Data regarding functional capacity, cardiopulmonary and vascular function post COVID-19 infection are scarce. To the best of our knowledge, few studies has evaluated functional capacity of patients recovering from COVID-19 infection and complications using cardiopulmonary exercise testing (CPET), and no study included endothelial function assessment.

Aims I. To investigate the effect of COVID-19 infection on cardiovascular and pulmonary function and exercise parameters in the pediatric and adult population.

II. To investigate the effect of PIMS on endothelial function in pediatric population.

Research hypothesis:

1. After COVID-19 infection, aerobic function is impaired due to cardiac and/or pulmonary limitation
2. Endothelial function in children after PIMS is impaired in comparison to healthy individuals and to patients after COVID infection with mild symptoms.

Importance of the study: Cardiovascular and pulmonary assessment of patients recovering from COVID-19 infection using CPET and Peripheral Arterial Tonography (EndoPAT™) has not been reported previously, and will provide new insights into the long term significance of COVID-19 infection.

DETAILED DESCRIPTION:
Introduction: coronavirus disease 2019 (COVID-19) pandemic caused by severe acute respiratory syndrome coronavirus 2 is currently a major public health challenge. COVID-19 infection results in diverse symptoms and morbidity. In severe cases, COVID-19 pathophysiology includes destruction of lung epithelial cells, thrombosis, and vascular leak leading to acute respiratory distress syndrome (ARDS) and subsequent pulmonary fibrosis. Clinical manifestations of COVID-19 can include cardiac involvement with complications, such as myocarditis (including fulminant cases), arrhythmias and rapid-onset heart failure. In children, severe acute infection is less common than in adults. Another COVID-19 related entity is a delayed life-threatening syndrome mimicking incomplete Kawasaki disease (KD) and toxic shock syndrome now designated as pediatric inflammatory multisystem syndrome (PIMS-TS) or MIS-C. Although rare, this syndrome remains an important source of pediatric COVID-19 related morbidity and mortality. The cardiovascular system is one of the major systems affected by this syndrome, manifesting mainly as myocarditis and/or coronary vasculitis. Endothelial dysfunction (ED) is a frequent long-term complication in patients after KD, manifesting as diminished production or availability of nitric oxide (NO) and an imbalance in the relative contribution of endothelium-derived relaxing and contracting factors. Little is known regarding ED post COVID-19 in the pediatric population but there is some evidence that endothelial injury might play a role in the pathogenesis of the disease. Patients who recover from acute COVID-19 infection or post-COVID-19 syndrome can have diverse complaints and symptoms such as chest pain, palpitations, weakness, myalgia and dyspnea. Several "return to play" guidelines exist for athletes, adults and children, due to concerns about long term cardiovascular and respiratory complications. Cardiopulmonary exercise testing (CPET) has become an important clinical tool to evaluate exercise capacity and predict outcome in patients with heart failure and other cardiac conditions. It provides assessment of integrative exercise responses involving the pulmonary, cardiovascular, and skeletal muscle systems, which are not adequately reflected through the measurement of individual organ system function. CPET is increasingly being used in a wide spectrum of clinical applications for evaluation of undiagnosed exercise intolerance and for objective determination of functional capacity and impairment. Few reports are available regarding CPET in post- COVID -19 infection adult patients, most of them after severe acute illness. Those reports demonstrated decreased aerobic capacity, not related to pulmonary limitation.

Peripheral Arterial Tonography (EndoPAT™) is a non-invasive and operator independent assessment of endothelial dysfunction. It evaluates the change in the volume of the pulse, using a volume sensor that is placed on the second fingertip both on the hand that is under evaluation and the free hand, measuring the reactive hyperemia mediated by NO release in response to local ischemia. EndoPAT™ has been in clinical research use for evaluation of endothelial changes in vasculitis, and has been deemed feasible and reproducible in the pediatric population. EndoPAT™, has been validated as a good evaluation tool for various blood-vessel related functions including arterial stiffness. In children, EndoPAT™ feasibility has been demonstrated in various conditions including inflammatory bowel disease (IBD) and Type I diabetes mellitus. We will therefore use this method to evaluate possible endothelial dysfunction in patients who suffered from PIMS. Endothelial dysfunction was previously evaluated by serum levels of endothelin, endothelin is a vasoconstricting substances that was previously used to evaluate endothelial dysfunction and high levels of endothelin were previously proved to be associated with coronary vasoconstriction. We aim to evaluate children, adolescents and adults, who had infection with COVID-19 or were diagnosed with PIMS and compare them to healthy controls, using pulmonary function tests, echocardiography, 6-min walk test (6MWT), CPET ,EndoPAT™ and serum levels of endothelin in order to identify long term cardiac or pulmonary residual function/limitation which might explain the symptoms or the long-term cardiopulmonary sequela of COVID-19 infection. Study design: Pediatric and adult patients recovering from COVID-19 with or without complaints or followed at the PIMS outpatient clinic or referred to the CPET clinic at Rambam Medical Center will be enrolled in the study. Data will be collected retrospectively/ prospectively, approximately 3 months after acute infection or post- COVID PIMS. CPET will be performed as part of the clinical evaluation recommended by the following physician. EndoPAT assesment- as part of the research. and blood endothelin levels- as part of the research. Participants will undergo all or part of the evaluation, and possibly repeated evaluations if needed. For CPET results each patient will be age- and sex-matched with an historical control from our CPET research database containing records of 200 healthy patients. For EndoPAT results- patient recovering from COVID-19 without PIMS will be evaluated as controls and the data will be compared to normal known values for age.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 5 years and older recovering from COVID-19 infection.
* For EndoPAT assessment-at least 3 months since the patient was diagnosed with COVID -19 infection or with PIMS

Exclusion Criteria:

* Cardiac or pulmonary comorbidity other than COVID-19 related morbidity.
* Inability to perform all study assessments. If a patient will be able to complete one of the assessments or more, the data will be collected and included in the analysis.
* Intercurrent systemic conditions or illness and/or medication use that could affect cardiopulmonary exercise capacity or EndoPAT™.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | Measured continuously during 15 minutes of the exercise test (CPET)
  Oxygen uptake evaluated by cardiopulmonary exercise testing (CPET)

SECONDARY OUTCOMES:
Six minute walk test (6MWT) | Six minutes
  patients will be instructed to walk as far as possible for six minutes in a 30-meter long enclosed corridor with a flat and hard surface, marked at every meter. Meters will be calculated at the end of the test.
Endothelin level | Five minutes for the blood to be drawn.
  One ml of serum will be needed using the Endothelin ELISA kit from R&D company.
Echocardiography | Ten minutes.
  Cardiac assessment using echocardiography for anatomical and functional evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel